CLINICAL TRIAL: NCT02047526
Title: A Non-interventional, Prospective Study to Evaluate the Clinical Epidemiology of Patients With Heart Failure (HF) in India
Brief Title: A Study to Evaluate the Clinical Epidemiology of Patients With Heart Failure (HF) in India
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-XXX-2012/1; HF Registry-India
Record Dates: First submitted 2013-02-06; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiovascular disease; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
This non-interventional, prospective, multi-centric, cross-sectional study is aimed to observe clinical practice in India in managing Heart Failure patients & to check one year outcome in HF patients. A total of 5 visits will be conducted during the study. There will be a baseline visit followed by four follow-up visits to assess the outcomes

DETAILED DESCRIPTION:
A non-interventional, prospective study to evaluate the clinical epidemiology of patients with Heart Failure (HF) in India

ELIGIBILITY:
Inclusion Criteria:

1. Provision of subject informed consent
2. Female or male aged 18 years and over
3. All patients with Dyspnea and/or signs of systemic congestion

Exclusion Criteria:

1. Subjects with Current Acute Coronary Syndrome
2. Absence of cardiac disease/structural heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Dyspnea and/or signs of systemic congestion
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular hospitalization rates and Length of stay | 1 year
HF related Hospitalization and hospital visits | 1 year
Cardiovascular and all cause mortality | 1 year
Change in Minnesota Living with Heart Failure Questionnaire scores. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Raza, MBBS, DIP DIAB, MBA, Study Director — AstraZeneca Pharma India Ltd.; R R Kasliwal, DM, Principal Investigator — Medanta, The Medicity, Gurgaon